CLINICAL TRIAL: NCT00823394
Title: African American Cancer Prevention Project: Establishing a Cohort to Investigate Health Disparities
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0970
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cancer
Keywords: African American; Adults; African American Cancer Prevention Project; Health Disparities; Questionnaire; Body Measurements; Self-help; Cancer Rates; Prevention
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires; Body Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Windsor Village United Methodist Church: Questionnaire + Body Measurements + Self-help Materials
  Interventions: Behavioral: Questionnaire; Other: Body Measurements; Behavioral: Self-help Materials

INTERVENTIONS:
Behavioral: Questionnaire — Completed privately via computer at Windsor Village Church, approximately 75 minutes. Repeated at Months 12 and 24.
  Other Names: Survey
Other: Body Measurements — Waist, hip, height, and weight measured privately. Repeated at Months 12 and 24.
Behavioral: Self-help Materials — Information on how to lower risk for developing cancer.

SUMMARY:
The goal of this research study is to learn if certain factors may affect cancer rates among African Americans. These factors include behavioral, social, and environmental factors including diet and physical activity, cigarette smoking, cancer screening, health care, neighborhood environment, and mental health.

DETAILED DESCRIPTION:
Study Procedures:

If you decide to take part in this study, you will complete study procedures at month 36 (the day you sign this consent form) and again every year for the next 2 years. These procedures include completing a questionnaire, having your body measurements taken, and receiving self-help materials.

At month 36, you will complete the questionnaire on a computer that is set up at the church in a private room. The questions will be about nutrition, exercise, tobacco and alcohol use, your neighborhood, age, education, social status, health status, stress, and racism. It should take about 75 minutes to complete. Your waist, hip, height, and weight will also be measured while you are in the private room.

Every year after that for the next 2 years, you will go back to the church to complete a new questionnaire each time. The questionnaires should take about 75 minutes to complete each time.

If you cannot get back to the church, you may complete the questionnaire over the phone. The study staff will provide you with the phone number and directions on how to complete the survey over the phone. Your measurements will be taken at the church, or at the Behavioral Research and Treatment Center (BRTC) at MD Anderson, whichever is more convenient for you.

At each study visit, you will also receive self-help materials on how to lower your risk for developing cancer.

Questionnaire Data:

Your questionnaire data will be used for research purposes only. Your responses will not be shared with your personal doctor. If you feel you need a doctor's opinion about anything that is asked about in the questionnaire (such as mental or emotional difficulties or symptoms), please contact your personal physician.

About 1 month after each you complete the questionnaire each time, the research staff will review and score your responses. If your scores suggest signs of depression, you will be given a list of resources for mental health screening.

Length of Study:

After 5 years, your active participation in this study will be over. You may be contacted in the future to see if you would agree to take part in other research studies.

This is an investigational study.

Up to 1,501 people will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. be age 18 years old and above
2. read and write English
3. live in the Houston metro area
4. have a viable (working) telephone number and home address

Exclusion Criteria:

1) None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult attendees of Windsor Village United Methodist Church living in Houston.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2008-12-05 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility Study Establishing African American Cancer Prevention Project (AACP) | 2 Years
  A longitudinal study to learn if and how certain behavioral, social, and environmental factors may affect cancer rates among African Americans as compared to other racial and ethnic groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna H. McNeill, MPH, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org